CLINICAL TRIAL: NCT06188065
Title: Associates of, and Time to Recovery From, Eosinopenia in Severe COPD Exacerbation
Brief Title: Eosinopenia in Severe COPD Exacerbation
Acronym: A-TREC
Status: Recruiting | Type: Observational
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: Newcastle University (Other); Chiesi UK (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SCI65
Record Dates: First submitted 2023-12-15; First posted 2024-01-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with severe exacerbation of COPD and eosinophils < 0.05 x 10^9/L: Participants to be included in the co-primary outcomes for the time to recovery from eosinopenia analysis as well as the analysis to identify independent factors associated with eosinopenia on admission in patients with a severe exacerbation of COPD. This group of participants will also be included in all secondary outcomes.
  Interventions: Diagnostic Test: Blood eosinophil count
- Participants with severe exacerbation of COPD and eosinophils >= 0.05 x 10^9/L: Participants will be included in the co-primary outcome to identify independent factors associated with eosinopenia on admission in patients with a severe exacerbation of COPD. This group of participants will also be included in some of the secondary outcomes.
  Interventions: Diagnostic Test: Blood eosinophil count

INTERVENTIONS:
Diagnostic Test: Blood eosinophil count — To determine the time it takes for blood eosinophil count to recover to baseline stable state following severe exacerbation of COPD associated with admission eosinopenia and to explore independent factors associated with admission eosinopenia.

SUMMARY:
The goals of this observational study are to identify factors independently associated with admission eosinopenia in patients with a severe exacerbation of chronic obstructive pulmonary disease (COPD) and to determine when blood eosinophil count (BEC) will recover to baseline stable state in patients who are admitted to hospital with a severe exacerbation of COPD and associated eosinopenia.

The main aims of the study are to:

1. Identify demographic, physiological and clinical factors independently associated with admission eosinopenia in patients with a severe exacerbation of COPD
2. Assess the time to recovery from eosinopenia to stable BEC following a severe exacerbation of COPD

DETAILED DESCRIPTION:
Blood eosinophils are a type of white blood cell that play a role in the immune system including fighting infection. They have numerous roles but are primarily involved in inflammation. They are recruited from the blood into sites of inflammation.

The blood eosinophil count (BEC) can be used as a biomarker to predict whether the addition of inhaled corticosteroid (ICS) to long-acting bronchodilators (LABD) will be beneficial in reducing future COPD exacerbations. This association is based on BEC being measured when patients are clinically stable. Patients with a higher BEC are more likely to gain these benefits where as conversely, patients with a lower BEC are less likely to benefit and the risk of side effects such as pneumonia will likely outweigh any potential benefit. Current national and international COPD guidelines suggest the use of BEC as a biomarker to help inform the decision of whether to commence or withdraw ICS, but do not specify measuring BEC at a time of clinical stability.

Decisions regarding changes to management are often made in the acute setting. Eosinophils transiently drop to very low levels in half of patients who are admitted to hospital with exacerbations of COPD. Measuring BEC during an acute illness risks incorrectly identifying all patients who may benefit from the introduction of an ICS. In the current BEC COPD study, reliance on admission and discharge BEC inappropriately denied ICS to 47% and 33% of patients respectively compared to a confirmed stable-state measure.

There are co-primary aims for this study. Firstly, the investigators wish to determine when BEC will recover to stable state following a hospital admission for exacerbation of COPD. Determining this will inform healthcare professionals of the optimum time to measure BEC for use as a biomarker when making decisions related to management escalation. Based on the results of BEC COPD, it is likely that an increased number of patients will be identified as being above the BEC threshold and therefore likely to benefit from ICS when time is allowed for BEC to recover to stable state. Appropriate introduction of ICS in this patient group will reduce exacerbation and hospital re-admission rates and thus may reduce overall mortality within this high-risk group. This should reduce the burden of COPD on patient's health, quality of life and the NHS.

Eosinopenia during severe exacerbation of COPD is associated with increased in-hospital and one year mortality. Treatment with oral corticosteroids does not fully explain the mechanism behind the development of eosinopenia, with the phenomenon being less common on discharge compared to admission despite inpatient oral corticosteroid treatment. The investigators other co-primary aim is to identify demographic, physiological and clinical factors independently associated with admission eosinopenia in patients with a severe exacerbation of COPD, providing useful mechanistic information regarding the relationship between BEC and short-term mortality.

The hypothesis for this study is that 90% of participants who are admitted to hospital with a severe exacerbation of COPD and eosinopenia will have recovery of their BEC to baseline stable state within 4 weeks. The investigators also hypothesize that there are demographic, physiological and clinical factors independently associated with admission eosinopenia other than prior systemic corticosteroid use.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital with primary clinical diagnosis of exacerbation of COPD*
* Smoking history of at least 10 pack years
* Airflow obstruction: FEV1/FVC ratio < 0.7 confirmed on historic or inpatient spirometry
* Capacity to give informed consent to participate

Exclusion Criteria:

* Parasitic infection, systemic fungal infection (excluding infection limited to nails or skin), eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome or other conditions associated with a high eosinophil count#
* Active malignancy
* Maintenance oral prednisolone or other systemic steroids, anti-interleukin 5 therapy or other medication known to influence eosinophils
* Patients with poor venous access
* Investigator confirmed history of asthma
* Non-COPD related health problems which in the view of the primary investigator may compromise the conduct and completion of the study

ADDITIONAL CRITERIA FOR THE TIME TO RECOVERY FROM EOSINOPENIA ANALYSIS ONLY

Inclusion criteria:

* Eosinopenia on admission
* Uneventful recovery*

  * Eosinopenia on admission who do not receive a further course of systemic corticosteroids or require emergency hospital admission for an acute illness in the six weeks following admission to hospital with a severe exacerbation of COPD.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be aged 35 years and over. They will have been admitted to hospital with an exacerbation of COPD +/- eosinopenia.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Indices independently associated with eosinopenia on admission in patients with a severe exacerbation of COPD. | On admission date
  Candidate indices will be identified by both univariate analysis (inclusion of indices related to eosinopenia at the 0.1 threshold) and domain knowledge (inclusion of indices thought likely to be related to eosinopenia even if no association on univariate analysis). Summary indices will also be created to reduce the number of variables (e.g. evidence of bacterial infection will include positive blood culture, sputum culture or antigens). Once candidate indices have been identifed, collinearity will be addressed and then independent associates of eosinopenia will be identified by logistic regression using backwards stepwise elimination.
The time taken for BEC to recover to stable state following a severe exacerbation of COPD. | 1, 2, 3, 4 and 6 weeks from admission date

SECONDARY OUTCOMES:
Level of agreement between the index admission eosinophil phenotype and prior admissions for exacerbations of COPD since May 2019. | On admission date
Change from baseline cytokine levels at day 28m stratified by intercurrent exacerbation or other acute illness status, including sub-group analysis (eosinopenic cohort vs non-eosinopenic cohort) | On admission date and 4 weeks from admission date
The proportion of patients whose BEC reaches 100 cell/uL or higher at each visit. | 1, 2, 3, 4 and 6 weeks from admission date
The time taken to reach peak BEC after a severe exacerbation of COPD. | 1, 2, 3, 4 and 6 weeks from admission date
Exploratory analysis looking for patient and treatment associations with rate of recovery of BEC. | 1, 2, 3, 4 and 6 weeks from admission date
  Patient and treatment variables associated with rate of recovery of BEC will be identified using univariate analysis.
Comparison of the rate of recovery of BEC in patients who had further exacerbations of COPD within the study period and patients who have not had further exacerbations. | 1, 2, 3, 4 and 6 weeks from admission date

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bourke, MBChB, PhD, Study Chair — Northumbria Healthcare NHS Foundation Trust; Peter Ireland, MBBS, Principal Investigator — Northumbria Healthcare NHS Foundation Trust
Locations (1):
- Northumbria Healthcare NHS Foundation Trust, North Shields, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bafadhel M, Peterson S, De Blas MA, Calverley PM, Rennard SI, Richter K, Fageras M. Predictors of exacerbation risk and response to budesonide in patients with chronic obstructive pulmonary disease: a post-hoc analysis of three randomised trials. Lancet Respir Med. 2018 Feb;6(2):117-126. doi: 10.1016/S2213-2600(18)30006-7. Epub 2018 Jan 10. PMID 29331313
- [Background] Singh D, Agusti A, Martinez FJ, Papi A, Pavord ID, Wedzicha JA, Vogelmeier CF, Halpin DMG. Blood Eosinophils and Chronic Obstructive Pulmonary Disease: A Global Initiative for Chronic Obstructive Lung Disease Science Committee 2022 Review. Am J Respir Crit Care Med. 2022 Jul 1;206(1):17-24. doi: 10.1164/rccm.202201-0209PP. No abstract available. PMID 35737975
- [Background] Suissa S, Ernst P. Precision Medicine Urgency: The Case of Inhaled Corticosteroids in COPD. Chest. 2017 Aug;152(2):227-231. doi: 10.1016/j.chest.2017.05.020. No abstract available. PMID 28797382
- [Background] Global Strategy for Prevention, Diagnosis and Management of COPD: 2023 Report. Global Initiative for Chronic Obstructive Lung Disease, 2023.
- [Background] Steer J, Gibson J, Bourke SC. The DECAF Score: predicting hospital mortality in exacerbations of chronic obstructive pulmonary disease. Thorax. 2012 Nov;67(11):970-6. doi: 10.1136/thoraxjnl-2012-202103. Epub 2012 Aug 15. PMID 22895999
- [Background] Prasad A, Echevarria C, Steer J, Bourke S C. Blood eosinophil counts during severe exacerbations do not reflect stable state inflammatory phenotype in COPD. European Respiratory Journal 2022 60: 1870.
- [Background] Lipson DA, Barnhart F, Brealey N, Brooks J, Criner GJ, Day NC, Dransfield MT, Halpin DMG, Han MK, Jones CE, Kilbride S, Lange P, Lomas DA, Martinez FJ, Singh D, Tabberer M, Wise RA, Pascoe SJ; IMPACT Investigators. Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD. N Engl J Med. 2018 May 3;378(18):1671-1680. doi: 10.1056/NEJMoa1713901. Epub 2018 Apr 18. PMID 29668352
- [Background] Lipson DA, Crim C, Criner GJ, Day NC, Dransfield MT, Halpin DMG, Han MK, Jones CE, Kilbride S, Lange P, Lomas DA, Lettis S, Manchester P, Martin N, Midwinter D, Morris A, Pascoe SJ, Singh D, Wise RA, Martinez FJ. Reduction in All-Cause Mortality with Fluticasone Furoate/Umeclidinium/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1508-1516. doi: 10.1164/rccm.201911-2207OC. PMID 32162970
- [Background] Echevarria C, Steer J, Prasad A, Quint JK, Bourke SC. Admission blood eosinophil count, inpatient death and death at 1 year in exacerbating patients with COPD. Thorax. 2023 Nov;78(11):1090-1096. doi: 10.1136/thorax-2022-219463. Epub 2023 Jul 24. PMID 37487711

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT06188065/Prot_SAP_000.pdf